CLINICAL TRIAL: NCT01580319
Title: Outpatient Strategy of Primary Prevention of Cardiovascular Diseases in Childhood and Adolescence: the Role of Physical Activity
Brief Title: Primary Prevention of Cardiovascular Diseases in Childhood and Adolescence: the Role of Physical Activity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in selecting the sample and follow-up lost.
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Principal Investigator, Claudia Ciceri Cesa, Master´s Degree, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2994/01
Record Dates: First submitted 2011-06-30; First posted 2012-04-19 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Obesity; Hypercholesterolemia; High Blood Pressure; Sedentary Lifestyle
Keywords: obesity; cholesterol; cholesterol, LDL; cholesterol, HDL; blood glucose; Triglyceride; C-Reactive Protein - hs; blood pressure; physical activity; Sedentary Lifestyle
MeSH Terms: conditions — Obesity; Hypercholesterolemia; Hypertension; Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants do not receive a physical exercise plan. Participants receive a simple orientations about lifestyle activities.
- Exercise (Experimental): Participants receive a physical exercise plan to play at home
  Interventions: Other: physical exercise

INTERVENTIONS:
Other: physical exercise — 150 minutes per week
  Other Names: physical activity; exercise
  Arms: Exercise

SUMMARY:
This research project is about a physical activity intervention in pediatric outpatients to try control and prevent heart diseases such as hypertension, obesity, high cholesterol.

DETAILED DESCRIPTION:
Control Group: receive information about health lifestyle Interventional Group: receive a structured plan with exercises to do 3 times per week within 50 minutes.

It is a randomized clinical trial and population are children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 17 years
* obesity
* high cholesterol

Exclusion Criteria:

* congenital heart diseases
* less than 6 or more than 17 years old

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Reduction on risk factors for a cardiovascular diseases (reduction on BMI, cholesterol, LDL, glucose, high-sensitivity C-reactive protein, blood pressure and/or increase on HDL) | These measurement were taken at end of followup (27th week)
  These measurement (taken at end of study) are assessed for a external research (blind for randomization) to judge the individual outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia C Cesa, MS, Principal Investigator — Instituto de Cardiologia
Locations (1):
- Instituto de Cardiologia / Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil